CLINICAL TRIAL: NCT01588340
Title: Comparison of Rapid Protocol Noncontrast MRI vs. Ultrasound in the Evaluation of Pediatric Hydronephrosis
Brief Title: MRI Hydronephrosis Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving institution
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jonathan R. Dillman M.D., Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: HUM00055762
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Hydronephrosis; Kidney Swelling
MeSH Terms: conditions — Hydronephrosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRI (Active Comparator): The patient will have a rapid noncontrast MRI (magnetic resonance imaging) that will take approximately 15 minutes to complete.
  Interventions: Procedure: MRI (Magnetic resonance imaging)
- Ultrasound exam (Active Comparator): A noncontrast ultrasound examination
  Interventions: Procedure: Ultrasound exam

INTERVENTIONS:
Procedure: MRI (Magnetic resonance imaging) — Subject will complete a 15 minute scan in the MRI
  Arms: MRI
Procedure: Ultrasound exam — The subject will complete a noncontrast ultrasound procedure that will take approximately 25 minutes to complete
  Arms: Ultrasound exam

SUMMARY:
The purpose of this study is to compare a rapid noncontrast MRI protocol not requiring sedation to ultrasound in the assessment of hydronephrosis.

DETAILED DESCRIPTION:
Ultrasound is the most commonly performed imaging modality used to assess hydronephrosis. The average renal ultrasound exam takes about 15-25 minutes to complete, however, it does have several disadvantages, including substantial operator dependence, having to rely on an adequate "sonographic window" to see the structures of interest and difficulty in visualization of portions of the kidney and urinary tracts.

Recent MRI advances have made rapid imaging possible. Such imaging has minimized motion related artifacts and need for sedation.

This study is to compare traditional ultrasound imaging to a raid noncontrast protocol MRI examination of the kidneys and urinary tract that would require no sedation and less than 15 minutes to perform.

ELIGIBILITY:
Inclusion Criteria:

* Children 2 years of age and younger
* Diagnosed with hydronephrosis and scheduled for an ultrasound scan

Exclusion Criteria:

* Healthy subjects

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2017-06 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
To assess the value of a rapid noncontrast MRI not requiring sedation to ultrasound in accurately diagnosing hydronephrosis in the pediatric patient. | 45 minutes
  A rapid MRI exam will be performed without IV contrast material or sedation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States